CLINICAL TRIAL: NCT05726617
Title: A Pilot Study : Avatar Intervention for the Treatment of Cannabis Use Disorder in Patients With Psychotic Disorders and/or Mood Disorders
Brief Title: Avatar Intervention for the Treatment of Cannabis Use Disorder in Patients With Severe Mental Health Disorders
Acronym: Avatar-CUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-12-2019-1564
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorders; Cannabis Use Disorder; Mental Health Disorder
Keywords: cannabis; virtual reality intervention; psychotic disorders; substance use disorders
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Marijuana Abuse; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: pilot clinical trial, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Avatar Intervention (Experimental): The Avatar Intervention will take place over 8 consecutive weeks, with one session per week. Each session will last approximately 60 minutes. The goal of the intervention will be to help you reduce cravings related to your cannabis use with the use of virtual reality and avatars.
  Interventions: Behavioral: Avatar Intervention

INTERVENTIONS:
Behavioral: Avatar Intervention — 8 weekly sessions of 60 minutes.
  Other Names: Avatar-CUD

SUMMARY:
This is a proof-of-concept of a new Virtual Reality (VR) Avatar Intervention for Cannabis Use Disorders (CUD) in patients with psychotic disorders and/or mood disorders. The primary outcomes are reductions in cannabis use, cannabis use disorder severity, and increased quality of life.

DETAILED DESCRIPTION:
Cannabis use disorder (CUD) is a complex issue, even more so when it is comorbid with a psychotic disorder or a mood disorder. Indeed, this population seems more vulnerable to this substance since the incidence of developing CUD is five to six times higher compared to the general population. In these populations, cannabis use is one of the key factors leading to psychiatric re-hospitalization. It is associated with depressive symptoms, medication non-compliance, hostility, as well as reduced quality of life. Unfortunately, there is no evidence-based intervention available for the treatment of CUD in this population. Novel interventions for CUD are thus critically needed. Virtual reality-based therapies are a promising avenue that allow patients to try novel strategies in real time instead of having to learn abstract concepts. In response to this clinical need, our team has created a distinctive intervention for CUD in patients with psychotic disorders and/or mood disorders. The Avatar Intervention displays strong experiential and relational components that are crucially missing in conventional interventions. This proposal thus aims to conduct a proof-of-concept to assess the efficacity of Avatar Intervention for CUD in patients with psychotic disorders and/or mood disorders. The primary objective of this open trial will be to determine whether cannabis-related outcomes (i.e. frequency and quantity of use) diminish after treatment as well as 3- 6- and 12-months follow-up. As for secondary objectives, the investigator will seek to determine the effect of the intervention on motivation to change, severity of cannabis dependence, psychiatric symptoms (mood and psychotic) and whether quality of life improves after treatment, at 3- 6- and 12-months follow-up. As there is no evidence-based therapeutic options for CUD in patients with psychotic disorders and/or mood disorders, the current trial will contribute to the validation of a novel approach and create new therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years of age who meet the DSM-5 criteria for CUD (≥4 criteria) ;
* Patients will meet the DSM-5 criteria for schizophrenia, schizoaffective disorder, bipolar disorder and major depression. Diagnoses will be established with the Structured Interview for DSM-5 (SCID-5).

Exclusion Criteria:

* Ongoing pharmacological or psychological treatment for CUD ;
* Ongoing detoxification for cannabis withdrawal ;
* Presence of neurological disorders ;
* Presence of a severe and unstable physical illness ;
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use (Timeline Follow-Back) | Within 1 week before treatment, within 1 week after treatment as well as 3- 6- and 12-months follow-up
  A standardized tool consisting of asking the patients how many joints they smoked each day of the week during the past week.

SECONDARY OUTCOMES:
Change in the severity of the cannabis use disorder (Cannabis Use Problems Identification Test - CUPIT) | Within 1 week before treatment, within 1 week after treatment as well as 3- 6- and 12-months follow-up
  16-item self-reported questionnaire assessing cannabis use and dependence; Range 3-82, higher values indicating a more severe cannabis use disorder
Change in quality of life (Quality of Life Scale -QLS) | Within 1 week before treatment, within 1 week after treatment as well as 3- 6- and 12-months follow-up
  QLS: 21-item scale based on a semistructured interview designed to assess deficit symptoms; Range 0-126, higher values indicate a better quality of life
Motivation to change cannabis use (Marijuana Ladder) | Within 1 week before treatment, within 1 week after treatment as well as 3- 6- and 12-months follow-up
  Diagram of a ladder with 10 "rungs," several of which are anchored by verbal labels of different degrees of readiness to change (pre-contemplation, contemplation, preparation, action, maintenance); higher values indicates a high degrees of readiness to change
Change in psychiatric symptoms (Positive And Negative Syndrome Scale - PANSS) | Within 1 week before treatment, within 1 week after treatment as well as 3- 6- and 12-months follow-up
  Positive And Negative Syndrome Scale: 30-item semi-structured interview investigating overall symptoms severity of schizophrenia in the last week; Subscales: Positive (7-49), Negative (7-49), General (16-112), Total score (subscales summed; 30-210); higher value indicates a worse symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, MD, PhD, Principal Investigator — University of Montreal, Institut universitaire en santé mentale de Montréal; Stéphane Potvin, PhD, Principal Investigator — University of Montreal, Institut universitaire en santé mentale de Montréal; Robert-Paul Juster, Study Chair — University of Montreal, Institut universitaire en santé mentale de Montréal
Locations (1):
- Research center of the Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No